CLINICAL TRIAL: NCT03668054
Title: Clinical Study for Evaluating the Safety and Clinical Effectiveness of Intravitreal Bevacizumab (Lumiere®) in Patients With Wet Age-related Macular Degeneration.
Brief Title: Safety and Clinical Effectiveness of Intravitreal Bevacizumab (Lumiere®) in Patients With Wet Age-related Macular Degeneration (Wet AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM2016
Record Dates: First submitted 2018-09-04; First posted 2018-09-12 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Open label, multicenter study for evaluating the safety and clinical effectiveness of intravitreal bevacizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab (Lumiere®) (Experimental): Dosage form: intravitreal single dose vial. Dosage: 0.05ml (1.25 mg) Frequency: monthly injections (up to 6 doses)
  Interventions: Drug: Bevacizumab (Lumiere®)

INTERVENTIONS:
Drug: Bevacizumab (Lumiere®) — The first three doses of bevacizumab (Lumiere®) were administered via intravitreal injection on a monthly basis. A safety evaluation was conducted in the first month. Following the first three doses, continuation of the treatment (up to 6 doses) was decided according to response.

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and clinical effectiveness of intravitreal bevacizumab (Lumiere®) in the single-dose form, for the treatment of patients with wet AMD.

DETAILED DESCRIPTION:
Age-related macular degeneration is the main cause of severe vision loss in patients over 65 years of age. There is solid evidence of the efficacy and safety of bevacizumab in the treatment of wet AMD. However, it has not been registered for such indication yet.

In response to the need for a proper adaptation, Lumiere® has been developed in a single-dose, sterile dosage containing bevacizumab 5 mg/vial in 0.2 mL injectable solution.

This adaptation is intended to assure intravitreal administration avoiding the risk of contamination and potential adverse consequences, such as endophthalmitis and blindness, associated to reutilization or repackaging of bevacizumab vials for oncological use.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years of age diagnosed with wet age-related macular degeneration having indication of antiangiogenic therapy.
* Both genders.
* Subjects able to give informed consent.

Exclusion Criteria:

* Patients with contraindication to receive bevacizumab:

  * Hypersensitivity to the active ingredient or to some of the formula excipients.
  * Hypersensitivity to products derived from CHO cells or to other human recombinant antibodies or humanized antibodies.
* Patients having received intravitreal antiangiogenic therapy prior to wet AMD treatment.
* Patients receiving previous systemic antiangiogenic therapy.
* Wet AMD in the healing period or disciform scar.
* Pregnant, breastfeeding or childbearing-aged women.
* Any person with choroidal neovascularization not associated to wet AMD.
* History of retinal or intraocular surgery in the affected eye in the last three months.
* Vitrectomy in the affected eye.
* Any significant ocular infection, active or suspected, having compromised or able to compromise the eye to be studied.
* Ocular inflammatory disease.
* Myopia exceeding -8 diopters.
* Extensive subfoveal subretinal hemorrhage > 2 papillary diameter (PD).
* Coexistence of other severe ocular diseases: uncontrolled ocular hypertension, terminal glaucoma, diabetic retinopathy, retinal vein thrombosis, optic atrophy.
* History of stroke or myocardial infarction in the last 6 months.
* Patients with coagulopathies.
* Patients physically or mentally disabled to participate in such visual tests.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events codified using MedDRA. | 6 months
  Register reports of drug related adverse events and compare them with prevalence in the literature after intravitreal bevacizumab (Lumiere®) in the single-dose form, for the treatment of patients with neovascular AMD.

SECONDARY OUTCOMES:
Number of participants with changes in visual acuity using the ETDRS charts in patients with wet AMD. | 6 months
Number of participants with changes in retinal thickness as assessed by OCT in patients with wet AMD. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Benisek, MD, Principal Investigator — Consultorios Médicos Dr. Benisek
Locations (3):
- Argentina (3):
  - Consultorios Médicos Dr. Benisek, Buenos Aires
  - Instituto Scorsetti S.A., Buenos Aires
  - Consultorios Médicos / Clínica de Cirugía Especializada S.A. (CCE), Buenos Aires

REFERENCES:
- [Result] Benisek DA, Manzitti J, Scorsetti D, Rousselot Ascarza AM, Ascarza AA, Gomez Rancano D, Quercia R, Ramirez Gismondi M, Carpio Total MA, Scorsetti ML, Spitzer E, Lombas C, Deprati M, Penna MI, Fernandez F, Tinelli MA. Safety and clinical effectiveness of intravitreal administration of bevacizumab (Lumiere(R)) in patients with neovascular age-related macular degeneration. Exp Ther Med. 2020 Dec;20(6):162. doi: 10.3892/etm.2020.9291. Epub 2020 Oct 9. PMID 33093900